CLINICAL TRIAL: NCT02106221
Title: Transforming Outcomes for Patients Through Medical Home Evaluation & reDesign
Acronym: TOPMED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Care Management Plus (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GBMF2908
Record Dates: First submitted 2014-03-21; First posted 2014-04-08 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Nurse Based Care Management; Health Information Technology
Keywords: Care coordination; nurse care management; practice facilitation; health information technology
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Financial incentives will be provided based on performance in areas determined to be of high-value.
  Interventions: Other: Intervention
- Control (Active Comparator): Financial incentives are a flat rate which can be reduced if an appropriate amount of effort or improvement is not met
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Will receive payments based on achievement in meeting goals based on specified high value elements as well as effort.
  Arms: Intervention
Other: Control — Will receive payments based on achievement in meeting goals.
  Arms: Control

SUMMARY:
The purpose of this study is to support enhancement, implementation, and evaluation of an improved model for delivering improved primary care to high-risk older adults through the use of health IT tools, focusing on issues related to the patient-centered primary care home (PCPCH) and other similar high-value elements that are proposed to improve patient outcomes. During this study, participating clinics will utilize the already-implemented Integrated Care Coordination Information System (ICCIS). Clinic staff will meet with a practice facilitator (monthly and as needed), and will track study activities and submit invoices via ICCIS reporting. These invoices will be used to simulate a shared savings model where clinics will be reimbursed based on their progress and effort towards their goals.

Clinics will set and work towards goals that they have chosen. Goals for the control arm are self-selected by the clinics themselves; goals for the invention arm are related to high-value elements (HVE) that have been identified as areas that can improve patient outcomes. These HVE are:

1. Evidence-based Care Management Based on Need
2. Identification of At-Risk Populations
3. Patient Engagement and Alerts Based on Goals
4. Integrated Information for Care Management, especially around Utilization
5. Population Management Tools

ELIGIBILITY:
Inclusion Criteria:

* clinics must be from the Oregon Rural Practice-based Research Network (ORPRN)
* Primary care clinic meeting one of the following health care setting descriptions: 1) small clinics in rural area, 2) medium-sized clinics in rural area, 3) clinics in moderate-sized health system, or 4) clinic within an academic medical center;
* Clinic will or has attested for PCPCH, achieving Tier 2 or 3 (of 3 tiers);
* Clinic is willing to contract to be a PCPCH with payers;
* Clinic has stable electronic health record (EHR) system with no plans to change systems during study duration;
* Clinic has willingness to receive practice facilitation and participate in study activities, including completion of assessments;
* Clinic has willingness to engage with research team members as defined in the study.

Exclusion Criteria:

* patients less then 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65500 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Preventable utilization | 12 months
  Reduce by 15% ED visits and hospitalizations related to ambulatory care
Quality Measures Improvement | 12 months
  Select 3 standard measures related to the patient population and improve each by 20%. (An example of such a measure might be fall risk assessment. There are several quality measures that are included as part of the HIT tool that is provided to clinics.)
Patient Satisfaction | 12 months
  Improve patient experience with clinic and satisfaction with care coordination by 10% Patient satisfaction will be determined by a CAHPS patient satisfaction survey that is sent out at the start and end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David A Dorr, MD, MS, Principal Investigator — Oregon Health and Science University; Marsha Pierre-Jacques Williams, BA, Study Chair — Oregon Health and Science University; Kimberley Gray, BSN, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Dorr DA, McConnell KJ, Williams MP, Gray KA, Wagner J, Fagnan LJ, Malcolm E. Study protocol: transforming outcomes for patients through medical home evaluation and redesign: a cluster randomized controlled trial to test high value elements for patient-centered medical homes versus quality improvement. Implement Sci. 2015 Jan 22;10:13. doi: 10.1186/s13012-015-0204-6. PMID 25609501